CLINICAL TRIAL: NCT06944834
Title: A Study on the Safety and Functionality of the Implantable Wireless Brain-Computer Interfaces for Motor Rehabilitation
Acronym: STAIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai StairMed Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PI2302-CL-01-002; JJ202503-01 (Other: IEC of Institution for National Drug Clinical Trials, Tangdu Hospital, Fourth Military Medical University)
Record Dates: First submitted 2025-04-08; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-03

CONDITIONS: Quadriplegia; Amputations; Spinal Cord Injuries (SCI); Brainstem Stroke
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries; Brain Stem Infarctions | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implantation of the WRS64 (Experimental): Implantation of the device and follow-up
  Interventions: Device: Implant

INTERVENTIONS:
Device: Implant — Implantation of the device and follow-up

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of minimally invasive, wireless brain-machine interface system (WRS) in patients with paralysis (resulting from spinal cord injuries, brainstem strokes, amyotrophic lateral sclerosis, or other motor neuron diseases causing complete or incomplete quadriplegia) or bilateral upper limb amputations. By leveraging brain-machine interface alternative technology, participants can use brain signals to control external devices (such as moving cursors, wheelchairs, robotic arms, WeChat Mini Programs, and other physical assistive devices), thereby improving their motor function and quality of life.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and efficacy of minimally invasive, wireless brain-machine interface system (WRS) in patients with paralysis (resulting from spinal cord injuries, brainstem strokes, amyotrophic lateral sclerosis, or other motor neuron diseases causing complete or incomplete quadriplegia) or bilateral upper limb amputations. By leveraging brain-machine interface alternative technology, participants can use brain signals to control external devices (such as moving cursors, wheelchairs, robotic arms, WeChat Mini Programs, and other physical assistive devices), thereby improving their motor function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years;
* Patients with complete or incomplete quadriplegia due to spinal cord injury, brainstem stroke, amyotrophic lateral sclerosis (ALS), or other motor neuron diseases, or those with bilateral upper limb amputations;
* Normal motor cortex function confirmed by neurological assessment;
* Muscle strength of bilateral or unilateral upper limbs ≤ Grade 3;
* Patients who have received standardized treatment and met diagnostic criteria for at least 12 months before screening, with stable disease status for ≥6 months;
* Expected lifespan ≥12 months;
* Normal cognitive function;
* Normal hearing and vision, or corrected vision to normal with standard lenses;
* Patients with stable caregivers;
* Willing to sign informed consent and able to comply with follow-up requirements.

Exclusion Criteria:

* Patients with neuropsychiatric disorders or psychological impairments;
* Patients with brain MRI findings showing hemorrhage, tumors, anatomical abnormalities, or distortions;
* History of severe systemic diseases (e.g., cardiac, pulmonary, hepatic, renal, thyroid, gastrointestinal, or hematologic disorders), poorly controlled diabetes, or pregnancy in females;
* History of infectious diseases (e.g., syphilis, HIV), severe traumatic brain injury, or major surgeries;
* Presence of metal implants or devices (e.g., cochlear implants, pacemakers, neurostimulators, defibrillators), except for dental implants or other implants deemed non-interfering;
* Surgical or anesthesia contraindications as determined by surgeons or anesthesiologists;
* Morbid obesity (BMI >40);
* Hearing impairment or uncorrectable visual deficits that would hinder prolonged computer monitor viewing;
* Current participation in other clinical trials;
* Other conditions considered unsuitable by investigators or medical staff.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Within 6 months after implantation
  The incidence of adverse events associated with the device or surgical procedure

SECONDARY OUTCOMES:
WRS Efficacy Assessment- Accuracy | 6 months after the implantation
  Validation of motor function improvement through cursor control performance metrics: the accuracy of of task list (number of correct items/ number of all items), the higher the better.
WRS Efficacy Assessment- Path efficiency | 6 months after the implantation
  Validation of motor function improvement is demonstrated through cursor control performance metrics, particularly path efficiency (the ratio of optimal to actual movement path). Higher values indicate better motor control performance.
WRS Efficacy Assessment- Time consumption | 6 months after the implantation
  Motor function improvement is validated through cursor control performance metrics, particularly time consumption (total task completion duration). Shorter durations indicate superior motor performance.
Neurological Recovery Assessment | 3, 15, 30, 90, 180 days after implantation
  The International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) scale was used to evaluate overall neurological status. The higher the scale score, the better the overall neurological status.
Changes in Quality of Life | 3, 15, 30, 90, 180 days after implantation
  Variations in the MOS item short from health survey (SF-36) scores were evaluated during both the main study period and long-term follow-up phase (comparing baseline to 6-month post-implantation assessments). The score values directly reflect health status - higher scores indicate better functional outcomes and superior quality of life.
Changes in Cognitive Performance | 3, 15, 30, 90, 180 days after implantation
  Variations in Montreal Cognitive Assessment (MoCA) scores scores were evaluated during both the main study period and long-term follow-up phase (comparing baseline to 6-month post-implantation assessments). Elevated scores are associated with improved cognitive function.
Changes in Psychological Status | 3, 15, 30, 90, 180 days after implantation
  Variations in Patient Health Questionnaire (PHQ-9) scores were evaluated during both the main study period and long-term follow-up phase (comparing baseline to 6-month post-implantation assessments). Higher scores indicate poorer psychological status.
Changes in Anxiety Status | 3, 15, 30, 90, 180 days after implantation
  Variations in Hamilton Anxiety Rating Scale (HAMA) scores were evaluated during both the main study period and long-term follow-up phase (comparing baseline to 6-month post-implantation assessments). Higher scores indicate poorer psychological status.
Changes in Depression Status | 3, 15, 30, 90, 180 days after implantation
  Variations in Hamilton Depression Rating Scale (HAMD) scores were evaluated during both the main study period and long-term follow-up phase (comparing baseline to 6-month post-implantation assessments). Higher scores indicate poorer psychological status.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No